CLINICAL TRIAL: NCT01204840
Title: Co-treatment With Recombinant Growth Hormone (GH) in Poor Responders Treated by in Vitro Fertilization (IVF-ET)
Brief Title: Growth Hormone for Poor Responders in in Vitro Fertilization (IVF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Fertility Centre (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Dr. Arthur Leader, Consultant, Ottawa Fertility Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OFC-001
Record Dates: First submitted 2010-09-14; First posted 2010-09-17 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Infertility; Poor Ovarian Reserve
Keywords: in vitro fertilization; IVF; poor responder; growth hormone; Poor responders to in vitro fertilization treatments
MeSH Terms: conditions — Infertility | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - Control group (Active Comparator): Group A (n=10; control group) will receive the "patch protocol" consisting of the 100ug estrogen patch (Estradot), a Gonadotropin Releasing Hormone (GnRH) antagonist (Cetrotide; 0.25mg/d), and gonadotropin stimulation with 412 IU of recombinant follicle stimulating hormone (r-FSH; Gonal F) and 150 IU of recombinant luteinizing hormone (r-LH; Luveris).
  Interventions: Drug: Patch protocol
- Group B - treatment group (Experimental): Group B will consist of 30 subjects. In addition to the same hormone stimulation "patch protocol" as Group A, subjects will be treated with growth hormone 10 IU (3.33mg) per day by subcutaneous injection starting day 1 of the last menstrual period in the month prior to gonadotropin stimulation, and will continue daily until the day of human chorionic gonadotropin (hCG) injection.
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — Subjects in this trial will use a 3.33mg vial (1 vial =10 IU) by daily subcutaneous injection. This will start on day 1 of the menstrual cycle preceding the stimulation phase of an IVF cycle, and will continue until the day of the human chorionic gonadotropin (hCG) trigger (approximately 5-6 weeks)
  Other Names: Saizen (Somatoptropin; Human growth hormone)
  Arms: Group B - treatment group
Drug: Patch protocol — Group A (n=10; control group) will receive "patch protocol": 100ug estrogen patch (Estradot), Gonadotropin releasing hormone (GnRH) antagonist (Cetrotide; 0.25mg/d), gonadotropin stimulation 412 IU recombinant follicle stimulating hormone (r-FSH; Gonal F) and 150 IU of recombinant luteinizing hormone (r-LH; Luveris). With 3 or more follicles at mean diameter equal to or greater than 17mm, urinary human chorionic gonadotropin (u-hCG) 10,000 IU self-injected to complete final maturation of oocytes. Egg retrieval will occur 36 hours after hCG injection. Eggs fertilized by standard IVF or intra-cytoplasmic sperm injection (ICSI) depending on semen parameters. Embryos cultured to day 2 and the best 2-4 will be transferred back under ultrasound guidance. Surplus embryos will be frozen as per clinic protocol. Luteal support: Endometrin 100mg vaginally three times daily, starting on the day of egg retrieval and continuing until menses or positive serum beta-hCG, then stopped.
  Arms: Group A - Control group

SUMMARY:
The purpose of this study is to determine if growth hormone given 4 weeks before as well as during a cycle of in vitro fertilization will improve outcomes in women who have had previous failure with IVF treatment cycles using high doses of follicle stimulating medications and had a poor response (less than 6 follicles).

DETAILED DESCRIPTION:
Growth hormone (GH; Saizen®) is indicated for the treatment of growth hormone deficiency in both children and adults, as well as for Turner's Syndrome, chronic renal failure, and children born short for gestational age.

In animal studies, growth hormone has been shown to be important in early antral follicle recruitment, subsequent follicular growth, and oocyte maturation. Together with insulin-like growth factor-1 (IGF-1), growth hormone is essential early on in the recruitment of primordial follicles in the growing pool (Slot et al 2006, Wandji et al 1992, Donadeu & Peterson 2008, Scaramuzi et al 2006, Liu et al, 1998).

Two recent meta-analyses have concluded that the addition of growth hormone during the ovarian stimulation phase of in vitro fertilization (IVF) cycles in poor responders will result in an increased probability of clinical pregnancy (Kolibianakas et al, 2009 and Ahmad et al, 2009). However, these studies have investigated the role of growth hormone in IVF when starting growth hormone injections with the initiation of gonadotropin stimulation. This may be too late to show an effect as GH may have more of an impact in the month prior to stimulation when primordial follicles are in the recruitment phase. Adding growth hormone in the month prior to stimulation with gonadotropins, as well as during stimulation phase may improve IVF outcomes by increasing the number of antral follicles that are recruited in the month prior to a stimulated cycle, and may ultimately improve the response to gonadotropin stimulation.

Starting growth hormone prior to stimulation has been studied in one previous publication (Kucuk et al, 2008), and showed that by starting growth hormone on day 21 of the menstrual cycle preceding gonadotropin stimulation, and continuing co-treatment with growth hormone until human chorionic gonadotropin (hCG) trigger resulted in a significantly higher number of fertilized oocytes when compared to a control group receiving no growth hormone (4.4 +/-1.8 vs 1.5 +/-0.9; p<0.001).

The addition of growth hormone to an IVF treatment protocol is directed at those infertile women who have previously undergone an IVF cycle on maximal doses of gonadotropins with a poor ovarian response. This study is aimed at improving IVF success in this population of women at the Ottawa Fertility Centre.

The purpose of this study is to determine if the addition of growth hormone both in the month prior to gonadotropin stimulation and during the active phase of stimulation, will result in an increased number of mature oocytes retrieved in previously poor responders during an IVF cycle.

ELIGIBILITY:
Inclusion Criteria:

* less than 42 years of age
* previous IVF cycle with high doses of gonadotropins (defined as greater than or equal to 400 IU/day)
* produced less than 6 follicles greater than or equal to 15mm

Exclusion Criteria:

* any known contraindications to the approved fertility drugs as per the Canadian Product Monographs
* any contraindications to growth hormone, pregnancy (to be ruled out and documented before GH treatment), or are at risk for gestational diabetes

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
number of mature oocytes retrieved | 8-12 weeks from IVF start date

SECONDARY OUTCOMES:
duration of stimulation | 8-12 weeks from IVF start date
gonadotropin requirements | 8-12 weeks from IVF start date
number of cumulus-oocyte complexes retrieved | 8-12 weeks from IVF start date
number of fertilized oocytes | 8-12 weeks from IVF start date
proportion of patients reaching embryo transfer | 8-12 weeks from IVF start date
implantation rate | 8-12 weeks from IVF start date
clinical pregnancy rate | 8-12 weeks from IVF start date

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Leader, BSc., MD, FRCSC, Principal Investigator — Ottawa Fertility Centre
Locations (1):
- Ottawa Fertililty Centre, Ottawa, Ontario, Canada

REFERENCES:
- See also: Ottawa Fertility Centre webpage — http://www.conceive.ca